CLINICAL TRIAL: NCT06877104
Title: Healing at Home 2.0 - Enhanced Chat Tool for Lowering Postpartum Depression
Acronym: HEALED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: March of Dimes (Other)
Responsible Party: Principal Investigator, Kirstin Leitner, Assistant Professor of Clinical Obstetrics and Gynecology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 857508
Record Dates: First submitted 2025-03-08; First posted 2025-03-14 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Depression, Postpartum; Postpartum Care
Keywords: Chat tool; Depression; Text message based program; Postpartum Care
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Routine postpartum care.
- Healing @ Home Program (H@H 2.0) (Experimental): Routine postpartum care and the use of an algorithm-based text message support program for six weeks.
  Interventions: Other: Healing @ Home Program (H@H 2.0)

INTERVENTIONS:
Other: Healing @ Home Program (H@H 2.0) — Healing @ Home 2.0 is a clinically used comprehensive technology-based postpartum support program, which provides 24/7 support to individuals through use of a text message based chatbot for six weeks postpartum. Content of H@H 2.0 includes anticipatory guidance regarding physical recovery, infant care and feeding, clinical algorithms to respond to urgent patient needs.
  Other Names: Penny the Chatbot; H@H 2.0; W2H
  Arms: Healing @ Home Program (H@H 2.0)

SUMMARY:
The purpose of the study is to determine if access to a text-message based holistic chatbot support program "Healing at Home 2.0" decreases depressive symptoms as measured by the Edinburgh Postnatal Depression Scale (EPDS) compared to usual postpartum care for patients of color.

DETAILED DESCRIPTION:
Healing at Home (H@H) 2.0 is a comprehensive technology-based postpartum support program which provides 24/7 support to individuals through use of an SMS chatbot for six weeks postpartum. This will be a randomized controlled trial (RCT) with an intervention arm consisting of patients who are planning to be discharged at routine timing (as determined by their clinical team) with access to H@H 2.0 postpartum SMS chatbot platform and a control arm which consists of usual postpartum care.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum patients who have delivered a singleton baby at or after 37w0d at the Hospital of the University of Pennsylvania
* Self-identify as a person of color (listed on chart as non-White race and confirmed with patient)
* Able to speak, read and write English
* Age ≥18
* Prenatal care at outpatient practice affiliated with the Hospital of the University of Pennsylvania
* Completion of clinically administered EPDS during inpatient stay
* Routine discharge timing, day 2 or more after vaginal delivery, day 3 or more after cesarean delivery

Exclusion Criteria:

* Unable to provide informed consent
* Baby not discharged with mother at postpartum discharge
* Does not have access to a mobile phone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 156 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) Screening Score | At 6 weeks postpartum
  Scores from the validated EPDS screening tool will be calculated using standard scoring criteria for each of the 10 items. A score of 9 or greater or indication of suicide ideation will be used to indicate a positive depression screen.

SECONDARY OUTCOMES:
Postpartum visit attendance | Up to 3 months postpartum
  Whether or not the patient attended their routine postpartum visit which should occur around the 6-week postpartum mark. We will accept routine postpartum visits up to 12-weeks postpartum.
Count of unscheduled emergency room/postpartum triage visits | Up to 6 weeks postpartum
  The number of unscheduled visits, reason for visit, whether or not patient was admitted to hospital in the first 6 weeks postpartum will be counted
Mode of feeding | At baseline and 6 weeks postpartum
  Patient asked mode of feeding at two time points. Options are exclusively breastfeeding, formula feeding only, or both breast and formula feeding.
Scores of self-efficacy in infant care | At baseline and at 6 weeks postpartum
  Scores from the validated Self-efficacy in the Nurturing Role (SENR) tool will be calculated using Likert scale scoring criteria for each of the 16 items. Negative items are reverse-scored such that higher scores on the items always reflect greater self-efficacy.
Knowledge of postpartum warning signs | At baseline and at 6 weeks postpartum
  Using a question from the Pregnancy Risk Assessment measure survey (PRAMS) to ask patients to identify warning signs of complications that can occur after birth
Score of Postpartum sleep: quality | At baseline and at 6 weeks postpartum
  One question Likert scale ranking quality of sleep from terrible to excellent.
Postpartum sleep: hours | At baseline and at 6 weeks postpartum
  Average number of hours slept in the past 7 days.
Postpartum pain score | 24 hours prior to discharge from hospital
  Scores from a 10-item question from the validated Brief Pain Inventory short form will be calculated using Likert scale scoring criteria with scores ranging from 0-100. Higher scores mean higher pain.
Social support and maternal functioning score | At 6 weeks postpartum
  Scores from the validated Barkin Index of Maternal Functioning tool will be calculated using Likert scale scoring criteria for each of the 20 questions. The total score ranges from 0 to 120, with a score of 120 representing perfect functioning.
Implementation outcome: Acceptability of Intervention Measure | At 6 weeks postpartum
  4-item Likert scale where scores can range from 4 to 20. High scores indicate higher acceptability. Given to the intervention group only.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Leitner, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No